CLINICAL TRIAL: NCT06247254
Title: Telehealth-Enhanced Assessment and Management After Stroke-Blood Pressure (TEAMS-BP)
Brief Title: Telehealth-Enhanced Assessment and Management
Acronym: TEAMS-BP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00114353; 2020C3-21070 (Other: PCORI)
Record Dates: First submitted 2024-01-22; First posted 2024-02-07 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Blood Pressure
Keywords: Hypertension; Stroke; Cardiovascular events
MeSH Terms: conditions — Hypertension; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive Tailored Telehealth Management (ITTM) (Experimental): ITTM is a novel adaptation of the Home Blood Pressure Telemonitoring and Case Management to Control Hypertension (HyperLink) model, based on the premise that patients have social and functional barriers to blood pressure management. In the ITTM arm, barriers to care are identified and addressed through Blood Pressure Care Plan messaging and referrals to needed resources. The ITTM intervention includes a tailored Blood Pressure Care Plan and health coaching contracted through INTERVENT. INTERVENT services may be reimbursed using Chronic Care Management (CCM) and Remote Patient Monitoring (RPM) insurance billing codes. Blood pressure monitors and wearable physical activity trackers will be provided to participants as part of the study.
  Interventions: Behavioral: Intensive Tailored Telehealth Management
- Intensive Clinic Management (ICM) (Other): ICM is based on the Stenting and Aggressive Medical Management for Preventing Recurrent Stroke in Intracranial Stenosis (SAMMPRIS) model and includes blood pressure management at in-person follow-up visits occurring every 2 months when systolic blood pressures are at target (i.e., < 130 mmHg), and monthly when systolic blood pressure is ≥ 130 mmHg. Participants will also receive low-touch health promotion messaging via text messaging, with reminders focused on medication adherence, healthy diet, and physical activity and a tailored Blood Pressure Care Plan for managing stroke recovery. Participants will be encouraged to monitor their blood pressure at home and record values in logs. Blood pressure monitors will be provided as part of the study.
  Interventions: Behavioral: Intensive Clinic Management

INTERVENTIONS:
Behavioral: Intensive Clinic Management — Blood pressure management at in-person follow-up visits occurring every 2 months when systolic blood pressures are at target (i.e., < 130 mmHg), and monthly when systolic blood pressure is ≥ 130 mmHg. Participants will also receive low-touch health promotion messaging via text messaging, with reminders focused on medication adherence, healthy diet, and physical activity and a tailored Blood Pressure Care Plan for managing stroke recovery. Participants will be encouraged to monitor their blood pressure at home and record values in logs.
  Other Names: ICM
  Arms: Intensive Clinic Management (ICM)
Behavioral: Intensive Tailored Telehealth Management — Tailored Blood Pressure Care Plan and health coaching contracted through INTERVENT.
  Other Names: ITTM
  Arms: Intensive Tailored Telehealth Management (ITTM)

SUMMARY:
TEAMS-BP is a Patient-Centered Outcomes Research Institute (PCORI)-funded trial under the Phased Large Awards for Comparative Effectiveness Research (PLACER) funding mechanism to evaluate two comprehensive and evidence-based strategies for managing blood pressure (BP) following stroke.

DETAILED DESCRIPTION:
Hypertension affects nearly half of the US population (46% of adults) and is the strongest risk factor for recurrent stroke. Prevalence in patients with ischemic or hemorrhagic stroke in the US varies by region (highest in the South) ranging from 70% to 82%, and is associated with greater risk of recurrent stroke, major cardiovascular events, and death. A vital question for stroke patients and caregivers is how to prevent a recurrent stroke and further adverse events. Multiple clinical trials have shown that lowering BP reduces the risk for cardiovascular disease and stroke. Few trials, however, included stroke patients with a focus on secondary prevention nor were representative of vulnerable populations. The former US Surgeon General recently published a Call to Action focused on BP with three goals: 1) make hypertension control a national priority; 2) ensure that communities support hypertension control; and 3) optimize patient care for hypertension control.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ischemic stroke defined as acute brain, spinal cord, or retinal infarction based on objective evidence on imaging (such as a focal area of restricted diffusion on Magnetic Resonance Imaging [MRI]) in a defined vascular distribution or clinical evidence of focal ischemic injury based on symptoms persisting > 24 hours; or spontaneous hemorrhagic stroke defined as a focal collection of blood within the brain parenchyma that is non-traumatic and identified by brain computed tomography (CT) or brain MRI
* Age ≥18 years
* Discharged directly home from acute care or inpatient rehabilitation
* At least one of the following: documented history of hypertension; self-reported history of hypertension; use of
* hypertension medications (either prescribed prior to stroke, administered during hospital stay, or prescribed at discharge)
* Systolic Blood Pressure ≥ 130 mmHg
* Able to read and understand English or Spanish,
* Have access to a functioning smartphone or tablet with cellular connectivity
* Willing to install and use a study-compatible physical activity monitoring application on their smartphone or tablet or smartphone or tablet of a qualifying caregiver
* Stated agreement to participate in either intervention to which they are assigned and attend all required study visits,
* Consent to receiving Short Message Service (SMS) required as part of the study interventions
* Consent to enrollment in Chronic Care Management required as part of the study interventions,
* Provision of a signed and dated informed consent form

Exclusion Criteria:

* Subdural hematoma or subarachnoid hemorrhage
* Current participation in another stroke clinical trial precluding dual enrollment
* Presence of terminal illness, such as cancer, that limits life expectancy to <1 year
* Diagnosis of end-stage renal disease defined as permanent kidney dysfunction requiring the use of hemodialysis or peritoneal dialysis
* Pregnancy, lactation or planning to become pregnant
* Late-stage Alzheimer's disease or related dementia
* Transitioned to a facility such as skilled nursing or long-term care prior to enrollment
* Mid upper arm circumference > 45 cm/17.7 inches or < 22 cm / 8.66 inches
* Missing values for Systolic Blood Pressure or Patient Activation Measure (PAM) score at baseline
* Any condition that in the opinion of the study investigator would preclude the participant from being able to safely participate in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Attaining the Target Systolic Blood Pressure of <130 mmHg | Month 6
  Systolic blood pressure will be calculated as the average of the second and third of 3 successive measures by the research coordinator according to standard protocols at 6 months (Study Visit 3).

SECONDARY OUTCOMES:
Change in Systolic Blood Pressure (SBP) at from baseline to 6 months post-stroke | Baseline to Month 6
  Defined as the systolic blood pressure at baseline (Visit 1) subtracted from the systolic blood pressure at 6 months (Visit 3). At both time points, systolic blood pressure will be calculated as the average of the second and third of 3 successive measures by the research coordinator according to standard protocols
Number of major adverse cardiovascular events (MACE) | Month 12
  Prevalence of major adverse cardiovascular events (MACE) - death or hospitalization from myocardial infarction, coronary heart disease, or stroke - within 1 year following randomization.
Change in Patient Activation Measured with the Patient Activation Measure (PAM) | Month 6
  Defined as the PAM Score at baseline (Visit 1) subtracted from the PAM Score at 6 months (Visit 3). The PAM is a validated 13-item patient-reported outcome measure (PROM) that measures skills and confidence to self-manage chronic disease. Response options for the 13 items are disagree strongly, disagree, agree, agree strongly with an interval-level scale from 0 to 100. To obtain the total PAM score, a propriety scoring algorithm will be used, with higher PAM scores indicating higher patient activation. Change in PAM will be analyzed as a continuous variable.

OTHER OUTCOMES:
Change in blood pressures following treatment | Month 3 to Month 12
  Change in blood pressures
Change in Cognitive function scores as assessed by the Montreal Cognitive Assessment (MoCA) scores | Baseline to Month 6, Baseline to Month 12
  Change in Cognitive function scores as assessed by the Montreal Cognitive Assessment (MoCA) score - The MoCA is a well-validated tool consisting of 30 items that screens for mild cognitive impairment, is more sensitive to changes than the Mini-Mental State Exam (MMSE) due to inclusion of more complex executive function items, and can be feasibly administered in stroke populations. Each of the domains (Visuospatial/Executive, Naming, Memory, Attention, Language, Abstraction, Delayed Recall, and Orientation) are scored separately and the scores are summed to obtain a total score that falls between 0 and 30. A score above 26 is considered normal. Change in MoCA scores from baseline to 12 months post-stroke will be assessed.
Change in (PROMIS) Patient-Reported Outcomes Measurement Information System Scores | Baseline to Month 6, Baseline to Month 12
  The PROMIS-10 is a series of 10 questions that assess physical function; higher scores indicate higher physical function.
Change in Modified Rankin Scale (mRS) Scores | Baseline to Month 6, Baseline to Month 12
  The most widely-used global disability scale covering the range of functional outcomes that is intuitive for patients and clinicians, has excellent validity and correlates with other patient-centered outcome scales. A single point change is clinically relevant. The mRS is a 5-question scale, with final scoring ranging from 0-5. Participants who are known to be deceased are assigned a score of 6, and deaths will be ascertained from the National Death Index.
Change in Medication Adherence | Baseline at 6 months,, Baseline to 12 months
  As assessed by the PROMIS Medication Adherence Scale (PMAS) is a 9-item, generic self-reported, medication-taking behavior scale, validated in kidney transplant patients.69-71 It has undergone rigorous development. Change in medication adherence will be assessed relative to
Patient Satisfaction Score | Month 6
  Participants rate their likelihood of recommending treatment from 0 (not at all likely) to 10 (extremely likely to recommend. To calculate the net promotor score, participants are classified as detractors (scores of 0 to 6), passives (scores of 7 to 8) and promoters (scores of 9 to 10). The net promotor score is then calculated as the difference in the proportion of promotors minus the proportion of detractors and ranges from -1 to 1.
Treatment Burden Score | Month 6
  The hypertension management burden questionnaire assesses degree of burden on 8 items representing the domains of the intervention (e.g., blood pressure monitoring, medication management, and physical activity). Item responses are on a Likert scale ranging from 0 (not burdensome at all) to 4 (extremely burdensome). Item scores are summed to generate a summary score ranging from 0-32.

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Bushnell, MD, Principal Investigator — Wake Forest University Health Sciences; Wayne Rosamond, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication - no end date
Access Criteria: Anyone who wishes to access the data